CLINICAL TRIAL: NCT02610725
Title: Online Yoga for Individuals With Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Director of Psychology, Dauten Family Center for Bipolar Treatment Innovation, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P001362
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Mood Disorders; Bipolar Disorder; Depression
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga class (Other): A 30 minute online Hatha yoga video intervention will be administered to participants.Participants will only participate in one yoga class and complete follow-up questionnaires.
  Interventions: Other: Hatha yoga

INTERVENTIONS:
Other: Hatha yoga — Participants will be shown a 30 minute video of a yoga class that they will be invited to follow along with.

SUMMARY:
We are seeking to understand the acceptability of an online yoga class for individuals with mood disorders. MoodNetwork members who are 18 years old or over who have experienced depression, mania, or hypomania are invited to participate. About 200 MoodNetwork participants will take part in this study.

DETAILED DESCRIPTION:
Yoga practitioners view yoga as a way to promote good physical and mental health, rather than as a treatment for poor health. This world view may be appealing to patients, especially those concerned with the stigma of conventional mental health treatment, or with the narrow focus on decreasing symptoms (instead of a broader focus on living to one's full potential) that defines much of conventional mental health treatment. Yoga classes are widely available and relatively inexpensive compared to other depression treatments. Yoga can be practiced at home with the aid of video recordings or books. We propose to examine the acceptability and feasibility of online yoga practice for individuals with depression, mania, or hypomania.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Over age 18
* Self-report of having experienced depression, mania, or hypomania in their lifetime

Exclusion Criteria:

* Any contraindication to exercise (e.g., pregnant, physical injuries or any other reason prohibiting exercise).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louisa G Sylvia, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Class
Started | 281
Completed | 75
Not Completed | 206
Not completed — Lost to Follow-up | 197
Not completed — self-reported contraindication | 9

BASELINE CHARACTERISTICS:
Population: Participants who consented and were not screened out for medical contraindications.
Arm/Group | Yoga Class
Number analyzed (Participants) | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.22 (13.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender : Male | 31
  Gender : Female | 238
  Gender : Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 235
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 227
  More than one race | 25
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Affect Scale
Description: The PANAS is a 20-item questionnaire that contains two 10-item subscales for positive and negative affect, respectively. The positive affect subscale assesses domains of excitement, enthusiasm, and attentiveness, whereas the negative subscale measures domains of distress, guilt, and irritability. Each subscale score can range from 10-50 where higher scores indicate greater levels of affect.
Time Frame: Pre- and post-intervention, 40 min
Population: 140 participants completed the PANAS at pre-intervention. 52 had valid data at post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Class
Number analyzed (Participants) | 140
units on a scale
  Positive Affect Pre-Intervention | 23.39 (7.95)
  Positive Affect Post-Intervention: number analyzed (Participants) | 52
  Positive Affect Post-Intervention | 25.38 (9.40)
  Negative Affect Pre-Intervention | 22.99 (8.83)
  Negative Affect Post-Intervention: number analyzed (Participants) | 52
  Negative Affect Post-Intervention | 15.21 (7.04)
Statistical Analysis 1: Comparison: Yoga Class; Paired-samples t-tests were used to analyze change in affect after participating in the yoga class. Analyses were conducted to measure changes in both positive affect and negative affect. This entry describes positive affect analysis; Test type: Superiority; p = 0.013, t-test, 2 sided; 51 degrees of freedom; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-3.73 to -0.46], Standard Deviation 0.81 — Means were analyzed in (pre-post) format. A negative mean here indicates an increase in positive affect
Statistical Analysis 2: Comparison: Yoga Class; Paired-samples t-tests were used to analyze change in affect after participating in the yoga class. Analyses were conducted to measure changes in both positive affect and negative affect. This entry describes negative affect analysis; Test type: Superiority; p < 0.001, t-test, 2 sided; 51 degrees of freedom; Mean Difference (Final Values) = 6.06, 95% CI 2-sided [4.10 to 8.02], Standard Error of Mean 0.98 — Means were analyzed in a (pre-post) format. A positive mean indicates a decrease in negative affect

2. Secondary Outcome: Feasibility/Acceptability Questionnaire
Description: This measure was developed for this study. It includes a Likert Scale item assessing how much participants liked the class (1 "Disliked it very much" to 10 "Liked it very much"). It also collects qualitative feedback on what they liked, disliked, as well as any other commentary. Quantitative data from Likert items are the secondary outcome reported.
Time Frame: Post-Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Class
Number analyzed (Participants) | 50
units on a scale | 7.40 (2.27)

3. Secondary Outcome: Adverse Event Questionnaire
Description: A free response survey asking for detail on any pain or injuries that may be relevant or related to the online yoga class
Time Frame: Post-Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Class
Number analyzed (Participants) | 50
Participants
  No reported pain or discomfort | 41
  Pain or discomfort as a result of participating | 4
  Limitations from previously existing conditions | 4
  Soreness unrelated to study intervention or health | 1

ADVERSE EVENTS:
Time Frame: 40 minutes
Arm/Group | Yoga Class
All-Cause Mortality (participants affected / at risk) | 0/281
Serious Adverse Events (participants affected / at risk) | 0/281
Other Adverse Events (participants affected / at risk) | 12/281
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yoga Class (N=281)
Pain or discomfort as a result of participation (Musculoskeletal and connective tissue disorders) | 6 — Any amount of pain or soreness associated breathing or stretching when following along with the yoga class.
Limitations from previously existing conditions (Musculoskeletal and connective tissue disorders) | 5 — Any pain or discomfort that is the product of exacerbating any previously existing medical conditions that were minor enough so as not to be deemed ineligible at consent
Soreness unrelated to study intervention or health (Musculoskeletal and connective tissue disorders) | 1 — Any pain or discomfort related to circumstances beyond the scope of study procedures or other health conditions

LIMITATIONS AND CAVEATS:
This study utilized a single online yoga class as a pilot to assess feasibility. Results may not fully reflect changes associated with long-term yoga practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02610725/Prot_SAP_000.pdf